CLINICAL TRIAL: NCT03965572
Title: Factors and Outcomes Associated With Use of Cabergoline Among Postpartum Women in Israel
Brief Title: Factors and Outcomes Associated With Postpartum Cabergoline Use
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laniado Hospital (Other)
Responsible Party: Principal Investigator, Dr. Sarit Kalfon, Principal Investigator, Laniado Hospital
Other Study IDs: 0017-19-LND
Record Dates: First submitted 2019-05-15; First posted 2019-05-29 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Lactation Suppressed; Cabergoline Adverse Reaction; Postpartum DVT; Postpartum Depression
Keywords: cabergoline, lactation, suppression, postpartum care
MeSH Terms: conditions — Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Postpartum women who requested cabergoline: A cohort of postpartum women, after a live birth, who request cabergoline for lactation suppression.
- Control group: An age-matched cohort of women after a live birth who have not requested cabergoline for lactation suppression.

SUMMARY:
Cabergoline is frequently being requested by many postpartum women with a live newborn to suppress lactation. The aim of the study is to investigate which women desire such an intervention, and what side effects they are experiencing.

DETAILED DESCRIPTION:
Cabergoline is a dopamine receptor agonist. Outside of the United States, it is occasionally used to suppress lactation, most commonly after a pregnancy loss or stillbirth. However, the investigators noted that the patient population in Israel has been requesting cabergoline for administration after healthy births, for immediate lactation suppression.

Use of cabergoline after delivery comes with many concerns. One primary concern is that this medication can increase the risk of venous thrombotic events, particularly during postpartum when thrombosis risk is already elevated. Secondly, it may have effects that alter mood, which are similarly concerning during a vulnerable period when postpartum depression and other mental health disorders are common.

Finally, of course, is the issue that so many women are requesting lactation suppression immediately after birth, and therefore will not accrue the neonatal and maternal benefits of lactation.

The investigators want to understand the characteristics, demographics and other factors that lead these women to make this choice, as well as assess their risk of medical and psychological adverse effects from cabergoline used in the postpartum period.

During this study, the investigators will not be prescribing cabergoline or in any way affecting its use. The study will be recruiting as subjects women who requested and received cabergoline prescriptions independently, as is common practice throughout the country.

The study will involve three questionnaires with these subjects: one in the hospital, after birth; one a week after birth; and one 6 weeks after birth. The questionnaires will involve medical history, a validated lactation questionnaire, as well as demographic data. All data will be held in a private, password-locked database.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women
* After a live birth
* Requesting cabergoline for lactation suppression

Exclusion Criteria:

* those who request cabergoline for lactation suppression after a stillbirth or pregnancy loss

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: We are studying the demographics, motivations, and outcomes of women who request cabergoline for lactation suppression following a live birth.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
Demographics of women requesting cabergoline | immediate postpartum
  Demographics parameter of women requesting cabergoline- age, number of children, profession. Data will be collected using questionnaire
Number of participants experiencing immediate treatment-related adverse events | immediate postpartum
  Adverse effects experienced by women taking cabergoline within few days after treatment will be recorded using questionnaire
Number of participants experiencing early treatment-related adverse events | 1 week postpartum
  Adverse effects experienced by women taking cabergoline within 1 week after treatment will be recorded using questionnaire with focus on thromboembolic events, and depression or mood changes.
Number of participants experiencing late treatment-related adverse events | six weeks postpartum
  Adverse effects experienced by women taking cabergoline within 6 weeks after treatment, will be recorded using questionnaire, with focus on thromboembolic events, and depression or mood changes.

SECONDARY OUTCOMES:
Motivations conducting participants to ask for a lactation suppression drug immediatly after giving birth | immediate postpartum
  Questionnaire assessing motivations expressed by women requesting cabergoline for lactation suppression postpartum, using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Kalfon, MD, Principal Investigator — Laniado Hospital
Locations (1):
- Laniado Hospital, The Betty Retter Mother & Baby Medical Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AlSaad D, ElSalem S, Abdulrouf PV, Thomas B, Alsaad T, Ahmed A, AlHail M. A retrospective drug use evaluation of cabergoline for lactation inhibition at a tertiary care teaching hospital in Qatar. Ther Clin Risk Manag. 2016 Feb 9;12:155-60. doi: 10.2147/TCRM.S96298. eCollection 2016. PMID 26929627
- [Background] Eidelman AI. Breastfeeding and the use of human milk: an analysis of the American Academy of Pediatrics 2012 Breastfeeding Policy Statement. Breastfeed Med. 2012 Oct;7(5):323-4. doi: 10.1089/bfm.2012.0067. Epub 2012 Sep 4. No abstract available. PMID 22946888
- [Background] Ben Natan M, Wiener A, Ben Haim Y. Women׳s intention to exclusively breast feed: The Israeli perspective. Midwifery. 2016 Mar;34:173-177. doi: 10.1016/j.midw.2015.11.013. Epub 2015 Nov 22. PMID 26652854
- [Background] McGuire TM. Drugs affecting milk supply during lactation. Aust Prescr. 2018 Feb;41(1):7-9. doi: 10.18773/austprescr.2018.002. Epub 2018 Feb 1. No abstract available. PMID 29507453
- [Background] Oladapo OT, Fawole B. Treatments for suppression of lactation. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD005937. doi: 10.1002/14651858.CD005937.pub3. PMID 22972088
- [Background] Senat MV, Sentilhes L, Battut A, Benhamou D, Bydlowski S, Chantry A, Deffieux X, Diers F, Doret M, Ducroux-Schouwey C, Fuchs F, Gascoin G, Lebot C, Marcellin L, Plu-Bureau G, Raccah-Tebeka B, Simon E, Breart G, Marpeau L. Postpartum practice: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians (CNGOF). Eur J Obstet Gynecol Reprod Biol. 2016 Jul;202:1-8. doi: 10.1016/j.ejogrb.2016.04.032. Epub 2016 Apr 29. PMID 27155443
- See also: Interim Report from Ministry of Health — http://www.health.gov.il/PublicationsFiles/mabat18072012.pdf
- See also: Breastfeeding basics: lactation suppression — http://www.breastfeedingbasics.com/articles/lactation-suppression